CLINICAL TRIAL: NCT00159133
Title: Prodrome-Based Early Intervention With Antipsychotics vs. Benzodiazepine in Patients With First-Episode Schizophrenia After One Year Maintenance Treatment Under Further Maintenance Treatment vs. Stepwise Discontinued Drugs
Brief Title: Prodrome-Based Early Intervention With Antipsychotics vs. Benzodiazepines in First-Episode Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government); German Research Network On Schizophrenia (Network); Janssen-Cilag Ltd. (Industry); University of Bonn (Other); Humboldt-Universität zu Berlin (Other); Ludwig-Maximilians - University of Munich (Other); University of Göttingen (Other); University of Cologne (Other); Mainz University (Other); University Hospital Tuebingen (Other); Universität Duisburg-Essen (Other); University of Mannheim (Other); University of Jena (Other); Martin-Luther-Universität Halle-Wittenberg (Other); RWTH Aachen University (Other); University of Wuerzburg (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01GI 9932 - P 2.2.2.2
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2008-01-30 (Estimated); Status verified 2008-01

CONDITIONS: Schizophrenia; Psychoses
Keywords: Schizophrenia; first episode; prodrome based early intervention; antipsychotics - benzodiazepine; maintenance treatment; drug discontinuation
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Early intervention with benzodiazepines in case of prodromal symptoms of an impending relapse
  Interventions: Drug: antipsychotics vs. Lorazepam (Drugs)
- 2 (Active Comparator): Early intervention with antipsychotics in case of prodromal symptoms of an impending relapse
  Interventions: Drug: antipsychotics vs. Lorazepam (Drugs)

INTERVENTIONS:
Drug: antipsychotics vs. Lorazepam (Drugs) — Early intervention with low-dose antipsychotics vs. lorazepam (up to 3 mg/day) in case of early warning signs of an impending relapse;

SUMMARY:
Prodrome based early intervention with an antipsychotic drug vs. benzodiazepine was applied in patients with first episode schizophrenia after one year neuroleptic maintenance treatment. Two groups of patients were followed over a period of 1 year: one further on under maintenance neuroleptic treatment, the other one after stepwise drug discontinuation.

DETAILED DESCRIPTION:
In case of early signs of a relapse prodrome based early intervention with an antipsychotic drug (Haloperidol, Risperidone and other) vs. benzodiazepine (Lorazepam) was applied in patients with first episode schizophrenia after one year neuroleptic maintenance treatment. Two groups of patients were followed over a period of 1 year: one further on under maintenance neuroleptic treatment (Haloperidol, Risperidone and other) , the other one after stepwise drug discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* First-episode in schizophrenia (according ICD-10 F20)
* Age between 18 and 55
* Informed consent
* One year neuroleptic maintenance treatment

Exclusion Criteria:

* Residence outside of the catchment area
* Legal reasons
* Insufficient knowledge of the german language
* Substance abuse or addiction
* Pregnancy
* Serious physical illness
* Organic brain disease
* Contraindication to neuroleptic treatment

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 71 (Estimated)
Dates: Start 2001-11; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
relapse rate | 1 year

SECONDARY OUTCOMES:
psychopathology | 1 year
social and cognitive functioning | 1 year
side-effects | 1 year
drop-out | 1 year
quality of life | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Gaebel, Professor, Study Chair — Department of Psychiatry and Psychotherapy, University of Düsseldorf, Rhineland State Clinics Düsseldorf, Bergische Landstraße 2, 40629 Düsseldorf
Locations (1):
- German Research Network on Schizophrenia, Department of Psychiatry and Psychotherapy at the Heinrich-Heine-University Düsseldorf, Düsseldorf, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Gaebel W, Moller HJ, Buchkremer G, Ohmann C, Riesbeck M, Wolwer W, Von Wilmsdorff M, Bottlender R, Klingberg S. Pharmacological long-term treatment strategies in first episode schizophrenia--study design and preliminary results of an ongoing RCT within the German Research Network on Schizophrenia. Eur Arch Psychiatry Clin Neurosci. 2004 Apr;254(2):129-40. doi: 10.1007/s00406-004-0509-y. PMID 15146342
- See also: Click here for more information about this study: Pharmacological long-term treatment strategies for relapse prevention in first episode schizophrenia — http://www.kompetenznetz-schizophrenie.de